CLINICAL TRIAL: NCT06942442
Title: A Phase II Trial of Tebentafusp in HLA-A*02:01 Positive Patients With Advanced Clear Cell Sarcoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sarcoma Alliance for Research through Collaboration (Other)
Collaborators: Royal Marsden NHS Foundation Trust (Other); Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SARC045
Record Dates: First submitted 2025-03-21; First posted 2025-04-24 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-10

CONDITIONS: HLA-A*0201 Positive Cells Present; Clear Cell Sarcoma (CCS)
Keywords: sarcoma; Tebentafusp; HLA-A*0201 Positive; HLA-A*02:01-negative; HMB-45+ clear cell sarcoma; Unresectable clear cell sarcoma; metastatic clear cell sarcoma
MeSH Terms: conditions — Sarcoma, Clear Cell; Sarcoma | interventions — tebentafusp

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tebentafusp (Experimental): Tebentafusp will be administered via IV infusion on Days 1, 8, and 15 of a 21-day cycle. Treatment on C1D1 will be 20mcg, treatment on C1D8 will be 30 mcg. After this initial dosing period, beginning at C1D15 and beyond, patients are eligible to receive the full dose of 68 mcg. This escalated dose administered at C1D15 will be the dose used for the remainder of the treatment period unless dose reduction is implemented for toxicity.
  Interventions: Drug: Tebentafusp
- Physician's choice arm (Active Comparator): Patients who are HLA-A*02:01-negative and ineligible to receive tebentafusp will be prospectively enrolled onto a separate study arm and treated with physicians' choice of treatment. They will also be radiographically assessed at the same schedule as patients treated with tebentafusp, if feasible, and kept on this treatment arm until progression of disease or unacceptable toxicity on the physicians' choice regimen.
  Interventions: Drug: Physician's Choice

INTERVENTIONS:
Drug: Physician's Choice — Patients who are HLA-A*02:01-negative and ineligible to receive tebentafusp will be prospectively enrolled onto a separate study arm and treated with physicians' choice of treatment. They will also be radiographically assessed at the same schedule as patients treated with tebentafusp, if feasible, and kept on this treatment arm until progression of disease or unacceptable toxicity on the physicians' choice regimen.
  Arms: Physician's choice arm
Drug: Tebentafusp — Patients who screen positive for HLA-A*02:01 and meet the eligibility requirements will be treated with weekly tebentafusp
  Arms: Tebentafusp

SUMMARY:
This is a multi-center, open label, phase II study of tebentafusp in patients with unresectable or metastatic clear cell sarcoma (CCS).

DETAILED DESCRIPTION:
This will be a multi-center, open label, phase II study of tebentafusp in patients with unresectable or metastatic CCS. Patients who screen positive for HLA-A*02:01 and meet the eligibility requirements will be treated with weekly tebentafusp. Radiographic assessment via CT or MR (where CT is not feasible or per the investigator's discretion) will occur at baseline and every subsequent 6 weeks through 48 weeks, and then every 9 weeks thereafter. Patients will be treated until progression of disease or unacceptable toxicity. All patients treated with tebentafusp will undergo mandatory research biopsies at baseline and on-treatment (week 6), if it is safe and feasible to do so. Serial peripheral blood samples for correlative analysis will be collected at baseline and at various time points on treatment.

Patients who are HLA-A*02:01-negative and ineligible to receive tebentafusp will be prospectively enrolled onto a separate study arm and treated with physicians' choice of treatment. They will also be radiographically assessed at the same schedule as patients treated with tebentafusp, if feasible, and kept on this treatment arm until progression of disease or unacceptable toxicity on the physicians' choice regimen.

ELIGIBILITY:
Inclusion Criteria

* Age 18 years
* Histologically confirmed diagnosis of HMB-45+ clear cell sarcoma which is unresectable and/or metastatic
* HLA-A*02:01 positive
* ECOG Performance Status of £ 2 at screening
* At least one site of measurable disease on CT/MRI scan as defined by RECIST v 1.1 criteria. Baseline imaging must be performed within 28 days of Cycle 1 Day 1 of study.
* Adequate organ function within 28 days of Day 1 of study defined as:
* Absolute Neutrophil Count (ANC) ≥ 1.5
* Platelets ≥ 75
* ALT and AST ≤ 2.5 x institutional upper limit of normal (ULN) or ≤ 5.0 x institutional ULN if considered due to tumor
* Alkaline phosphatase ≤ 2.5 x institutional ULN unless considered due to tumor
* Serum bilirubin ≤ 1.5 x institutional ULN. NOTE: Patients with elevated bilirubin secondary to Gilbert's disease are eligible to participate in the study
* Serum creatinine ≤ 1.5 x institutional ULN or 24-hour creatinine clearance ≥ 50 ml/min (calculated creatinine clearance using Cockroft formula is acceptable)
* Written, voluntary informed consent
* Patients must demonstrate progression of disease by RECIST 1.1 within 6 months of study enrollment. Newly diagnosed patients with unresectable or metastatic disease and only one baseline scan are eligible to screen and enroll.
* All other relevant medical conditions must be well-managed and stable, in the opinion of the investigator, for at least 28 days prior to first administration of study drug

Exclusion Criteria:

* History of sever hypersensitivity reaction (e.g. anaphylaxis) to other biologic drugs or monoclonal antibodies
* Clinically significant cardiac disease or impaired cardiac function, including any of the following:
* Clinically significant and/or uncontrolled heart disease such as congestive heart failure (New York Heart Association grade ≥ 2), uncontrolled hypertension, or clinically significant arrhythmia currently requiring medical treatment
* QTcF > 470 msec on screening electrocardiogram (ECG) or congenital long QT syndrome. NOTE: If the initial automated QTcF interval is > 470 msec at screening, for the purpose of determining eligibility, the mean QTcF, based on at least 3 ECGs obtained over a brief time interval (ie, within 30 minutes), should be manually determined by a medically qualified person.
* Acute myocardial infarction or unstable angina pectoris < 6 months prior to Screening
* Presence of symptomatic or untreated central nervous system (CNS) metastases, or CNS metastases that require doses of corticosteroids within the prior 3 weeks to study Day 1. Patients with brain metastases are eligible if lesions have been treated with localized therapy and there is no evidence of progression for at least 4 weeks by MRI prior to the first dose of study drug
* Active infection requiring systemic antibiotic therapy. Patients requiring systemic antibiotics for infection must have completed therapy at least 1 week prior to the first dose of study drug
* Known history of uncontrolled human immunodeficiency virus (HIV) infection (defined as CD4 count < 200 and/or a detectable viral load). Testing for HIV status is not necessary unless clinically indicated
* Active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection per institutional protocol. Testing for HBV or HCV status is not necessary unless clinically indicated or the patient has a history of HBV or HCV infection
* Malignant disease, other than that being treated in this study. Exceptions to this exclusion include the following: malignancies that were treated curatively and have not recurred within 2 years prior to study treatment; completely resected basal cell and squamous cell skin cancers; any malignancy considered to be indolent and that has never required therapy; and completely resected carcinoma in situ of any type
* Any medical condition that would, in the investigator's or Sponsor's judgment, prevent the patient's participation in the clinical study due to safety concerns, compliance with clinical study procedures or interpretation of study results
* Patients receiving systemic steroid therapy or any other immunosuppressive medication at any dose level, as these may interfere with the mechanism of action of study treatment. Local steroid therapies (e.g., otic, ophthalmic, intra-articular or inhaled medications) are acceptable
* History of adrenal insufficiency
* Participants with clinically significant pulmonary disease or impaired lung function, including any of the following:
* An oxygen saturation of < 92% on room air, measured by pulse oximeter
* History of interstitial lung disease
* History of pneumonitis that required corticosteroid treatment or current pneumonitis
* Ongoing requirement for intermittent or continuous oxygen supplementation
* History of colitis or inflammatory bowel disease
* Major surgery within 2 weeks of the first dose of study drug (minimally invasive procedures such as bronchoscopy, tumor biopsy, insertion of a central venous access device, and insertion of a feeding tube are not considered major surgery and are not exclusionary)
* Radiotherapy within 2 weeks of the first dose of study drug, with the exception of palliative radiotherapy to a limited field, such as for the treatment of bone pain or a focally painful tumor mass
* Use of hematopoietic colony-stimulating growth factors (eg, G-CSF, GM- CSF, M-CSF) ≤ 2 weeks prior to start of study drug. An erythroid-stimulating agent is allowed as long as it was initiated at least 2 weeks prior to the first dose of study treatment and the patient is not red blood cell transfusion dependent
* Women who are pregnant or nursing/breastfeeding. Where pregnancy is defined as the state of a female after conception and until the termination of gestation.
* Women of childbearing potential who are sexually active with a non- sterilized male partner, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective contraception during study treatment (defined in Section 7.2.3), and must agree to continue using such precautions for 6 months after the final dose of investigational product: cessation of birth control after this point should be discussed with a responsible physician.
* Male patients must be surgically sterile or use double barrier contraception methods from enrollment through treatment and for 6 months following administration of the last dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2025-10-22 (Actual); Primary Completion 2030-10-01 (Estimated); Study Completion 2030-10-01 (Estimated)

PRIMARY OUTCOMES:
Measure Disease Response | Approximately 5.5 months
  To estimate the population of HLA-A*02:01-positive patients with metastatic or unresectable clear cell sarcoma and treated with tebentafusp who are progression free at 24 weeks. PFS (progression-free survival) will be determined using iRECIST.

SECONDARY OUTCOMES:
Progression-Free Survival | Approximately 5 years
  To determine the PFS, in this population at months 3 and 5. Progression-free survival (PFS) defined as the time from study entry to disease relapse, disease progression, or death from any cause, using iRECIST. Patients without an event will be censored at the time of last disease follow-up.
Estimate Overall Survival | Approximately 5 years
  To estimate the overall survival (OS) in patients who are HLA-A*02:01-positive with metastatic or unresectable clear cell sarcoma and treated with tebentafusp. Overall survival, defined as the time from study entry to death from any cause. Patients who are alive at the time of analysis will be censored at the date of last follow-up.
Objective Response Rate | Approximately 5 years
  To estimate the objective response rate (ORR) in patients who are HLA-A*02:01-positive with metastatic or unresectable clear cell sarcoma and treated with tebentafusp, according to iRECIST. Objective tumor response, defined as achievement of nadir response of complete response (CR) or partial response (PR) by iRECIST without prior progression any time during protocol therapy.
Duration of Response | Approximately 5 years
  To estimate the duration of response (DoR) in this population. DoR can be defined as the measurement of time from the start of treatment response to disease progression or death

OTHER OUTCOMES:
Progression-Free Survival and Objective Response Rate | Approximately 5 years
  To compare the 5-month PFS rate and ORR for patients who are HLA-A*02:01-positive with metastatic or unresectable clear cell sarcoma and treated with tebentafusp against patients who are HLA-A*02:01-negative with metastatic or unresectable clear cell sarcoma, according to RECIST 1.1. Duration of response is defined as the time from a nadir tumor response of CR/PR to disease progression.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Southern California - Norris Cancer Center, Los Angeles, California
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: No